CLINICAL TRIAL: NCT00369122
Title: A PHASE II STUDY OF BEVACIZUMAB IN COMBINATION WITH DEFINITIVE RADIOTHERAPY AND CISPLATIN CHEMOTHERAPY IN UNTREATED PATIENTS WITH LOCALLY ADVANCED CERVICAL CARCINOMA
Brief Title: Bevacizumab, Radiation Therapy, and Cisplatin in Treating Patients With Previously Untreated Locally Advanced Cervical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Radiation Therapy Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00722; NCI-2009-00722 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000493005; RTOG 0417 (Other: Radiation Therapy Oncology Group); RTOG-0417 (Other: CTEP); U10CA021661 (NIH); NCT01530633 (obsolete NCT alias)
Record Dates: First submitted 2006-08-24; First posted 2006-08-29 (Estimated); Results first posted 2013-05-17 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2018-02

CONDITIONS: Cervical Adenocarcinoma; Cervical Adenosquamous Carcinoma; Cervical Squamous Cell Carcinoma, Not Otherwise Specified; Stage IB Cervical Cancer AJCC v6 and v7; Stage IIA Cervical Cancer AJCC v7; Stage IIB Cervical Cancer AJCC v6 and v7; Stage III Cervical Cancer AJCC v6 and v7
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Brachytherapy

ARMS (1):
- Treatment (radiation therapy, bevacizumab, cisplatin) (Experimental): Patients undergo pelvic EBRT once daily, 5 days a week, for 5 weeks for a total of 45 Gy.
  Some patients also undergo low-dose rate brachytherapy twice, 1-3 weeks apart, beginning >= 4 weeks after initiating EBRT or high-dose rate brachytherapy 5 times, >= 48 hours apart, beginning >= 2 weeks after initiating EBRT. EBRT and chemotherapy are halted on the day of high-dose rate brachytherapy. Patients receive bevacizumab IV over 30-90 minutes on days 1, 15, and 29 and cisplatin IV over 60 minutes on days 1, 8, 15, 22, 29, and 35.
  Interventions: Biological: Bevacizumab; Drug: Cisplatin; Radiation: External Beam Radiation Therapy; Radiation: Internal Radiation Therapy

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar FKB238; BEVACIZUMAB, LICENSE HOLDER UNSPECIFIED; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Radiation: External Beam Radiation Therapy — Undergo EBRT
  Other Names: Definitive Radiation Therapy; EBRT; External Beam Radiotherapy; External Beam RT; external radiation; External Radiation Therapy; external-beam radiation
Radiation: Internal Radiation Therapy — Undergo brachytherapy
  Other Names: BRACHYTHERAPY; internal radiation; Internal Radiation Brachytherapy; Radiation Brachytherapy

SUMMARY:
This phase II trial is studying how well giving bevacizumab together with radiation therapy and cisplatin works in treating patients with previously untreated locally advanced cervical cancer. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of cervical cancer by blocking blood flow to the tumor. Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving bevacizumab together with radiation therapy and cisplatin may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine treatment-related serious adverse-event rates and adverse-event rates within the first 90 days from treatment start in patients with previously untreated locally advanced carcinoma of the cervix treated with bevacizumab, cisplatin, and concurrent pelvic radiotherapy.

SECONDARY OBJECTIVES:

I. Evaluate treatment-related serious adverse events and adverse events at any time.

II. Evaluate disease-free survival (local, regional, or distant failure, or death due to any cause).

III. Evaluate overall survival (death due to any cause). IV. Implement the image-based brachytherapy guidelines proposed by the Transatlantic Image-Guided Brachytherapy Working Group.

V. Collect CT scan or MRI-based dosimetry of brachytherapy applications used during the course of treatment for later analysis of feasibility and consistency as well as dose/volume assessments of tumor control and complications.

OUTLINE: This is a multicenter study.

Patients undergo pelvic external-beam radiotherapy (EBRT) once daily, 5 days a week, for 5 weeks for a total of 45 Gy.

Some patients also undergo low-dose rate brachytherapy twice, 1-3 weeks apart, beginning >= 4 weeks after initiating EBRT or high-dose rate brachytherapy 5 times, >= 48 hours apart, beginning >= 2 weeks after initiating EBRT. EBRT and chemotherapy are halted on the day of high-dose rate brachytherapy. Patients receive bevacizumab IV over 30-90 minutes on days 1, 15, and 29 and cisplatin IV over 60 minutes on days 1, 8, 15, 22, 29, and 35.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed squamous cell, adenocarcinoma, or adenosquamous cell carcinoma of the uterine cervix, meeting 1 of the following stage criteria:

  * Stage IIB-IIIB lymph nodes
  * Stage IB-IIA disease with biopsy-proven pelvic node metastases and/or tumor size >= 5 cm
* No positive para-aortic lymph nodes
* Zubrod performance status 0-2
* WBC >= 3,000/mm^3
* Absolute granulocyte count >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* INR < 1.5
* Total bilirubin =< 1.5 mg/dL
* Serum creatinine =< 1.5 mg/dL
* AST and ALT =< 2.5 times upper limit of normal (ULN)
* Serum calcium =< 1.3 times ULN
* Hemoglobin >= 10 g/dL (transfusion allowed)
* Urine protein:creatinine ratio ? 0.5 OR urine protein < 1,000 mg by 24-hour urine collection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* None of the following illnesses or conditions:

  * Medical illness preventing the use of full-dose chemotherapy
  * Evidence of bleeding diathesis or coagulopathy
  * Prior medical or psychiatric illness that would prevent informed consent or limit survival to < 6 months
  * History of aneurysms, cerebrovascular accident, or arteriovenous malformations
  * Active gastrointestinal (GI) ulcers, GI bleeding, or active inflammatory bowel disease
  * Serious, nonhealing wound, ulcer, or current healing fracture
  * History of any type of fistula or GI perforation
  * Intra-abdominal abscess within the past 6 months
* No prior invasive malignancy (except nonmelanomatous skin cancer) unless disease free for >= 3 years
* No significant traumatic injury within the past 28 days
* No clinically significant cardiovascular disease, such as the following:

  * Uncontrolled hypertension (blood pressure > 160/90 mm Hg on medication)
  * Myocardial infarction within the past 12 months
  * Unstable angina within the past 12 months
  * New York Heart Association class II-IV congestive heart failure
  * Unstable symptomatic arrhythmia requiring medication (i.e., chronic atrial arrhythmia, atrial fibrillation, or paroxysmal supraventricular tachycardia)
  * Arterial thromboembolic events, including transient ischemic attack or clinically significant peripheral artery disease, within the past 6 months
* Arterial thromboembolic events, including transient ischemic attack or clinically significant peripheral artery disease, within the past 6 months
* No known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* No known HIV
* No prior organ transplant
* No prior surgery for carcinoma of the cervix other than biopsy
* No prior surgical debulking of pelvic or para-aortic nodes
* No prior pelvic radiotherapy, including transvaginal irradiation to control bleeding
* No prior systemic chemotherapy
* No major surgical procedure or open biopsy within the past 28 days or anticipation of need for major surgical procedure during the course of the study
* No fine needle aspirations or core biopsies within the past 7 days
* No concurrent major surgical procedure
* No concurrent epoetin alfa or Hypericum perforatum (St. John's wort)
* No concurrent intensity-modulated radiotherapy
* No concurrent transvaginal irradiation to control bleeding

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-08-11 (Actual); Primary Completion 2010-06-04 (Actual); Study Completion 2016-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracey Schefter, Principal Investigator — Radiation Therapy Oncology Group
Locations (106):
- United States (103):
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - University of Colorado, Denver, Colorado
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Integrated Community Oncology Network-Southside Cancer Center, Jacksonville, Florida
  - University of Florida Health Science Center - Jacksonville, Jacksonville, Florida
  - Baptist Medical Center South, Jacksonville, Florida
  - Integrated Community Oncology Network-Florida Cancer Center Beaches, Jacksonville Beach, Florida
  - 21st Century Oncology-Orange Park, Orange Park, Florida
  - UF Cancer Center at Orlando Health, Orlando, Florida
  - 21st Century Oncology-Palatka, Palatka, Florida
  - Bay Medical Center, Panama City, Florida
  - Integrated Community Oncology Network-Flager Cancer Center, Saint Augustine, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Franciscan St. James Health-Olympia Fields Campus, Olympia Fields, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Saint Vincent Anderson Regional Hospital/Cancer Center, Anderson, Indiana
  - Franciscan Saint Francis Health-Beech Grove, Beech Grove, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Reid Health, Richmond, Indiana
  - Providence Medical Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Radiation Oncology Practice Corporation Southwest, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Shawnee Mission Medical Center-KCCC, Shawnee Mission, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - Norton Suburban Hospital and Medical Campus, Louisville, Kentucky
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Cape Radiation Oncology, Cape Girardeau, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Radiation Oncology Practice Corporation South, Kansas City, Missouri
  - Saint Joseph Health Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Radiation Oncology Practice Corporation - North, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - CHI Health Good Samaritan, Kearney, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - New York-Presbyterian/Brooklyn Methodist Hospital, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Highland Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Summa Barberton Hospital, Barberton, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Veteran Affairs Medical Center, Dayton, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Cancer Care Center, Incorporated, Salem, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Einstein Medical Center Philadelphia, Philadelphia, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Main Line Health NCORP, Wynnewood, Pennsylvania
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - M D Anderson Cancer Center, Houston, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Cottonwood Hospital Medical Center, Murray, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Intermountain Health Care, Salt Lake City, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - Southwest VA Regional Cancer Center, Norton, Virginia
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (3):
  - London Regional Cancer Program, London, Ontario
  - McGill University Department of Oncology, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Radiation Therapy, Bevacizumab, Cisplatin)
Started | 60
Completed | 49 (Subjects contributing data to the primary analysis are considered to have completed the study.)
Not Completed | 11
Not completed — Ineligible | 10
Not completed — No protocol treatment | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Radiation Therapy, Bevacizumab, Cisplatin)
Number analyzed (Participants) | 60
Age, Continuous [Median (Full Range); unit: years] | 45.5 [20 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Treatment-related Serious Adverse Events (SAEs) and Adverse Events (AEs) as Assessed by CTCAE v. 3.0 Criteria Within the First 90 Days From Treatment Start.
Description: Adverse events (AEs) graded using CTCAE v3.0. Grade (Gr) refers to the severity of the AE and assigns Gr 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: 1= Mild AE, 2= Moderate AE, 3= Severe AE, 4= Life-threatening or disabling AE, 5= Death related to AE. Treatment-related SAEs defined as Grade (Gr) >= 4 vaginal bleeding, Gr >=4 thrombotic event, Gr >=3 arterial event, gastrointestinal (GI) bleeding , or bowel/bladder perforation, and any Gr 5 treatment-related AE. Treatment-related AEs defined as all SAEs, Gr 3-4 nausea, vomiting, or diarrhea persisting for >2 weeks despite medical intervention, Gr 4 neutropenia or leukopenia persisting for >7 days, febrile neutropenia defined as a temperature >38.5 degree Celsius and granulocytes < 1000/mm3, Grade 3-4 hematologic toxicity with the exception of neutropenia and leukopenia, and Grade 3-4 GI, renal, cardiac, pulmonary, hepatic, or neurologic AEs.
Time Frame: From start of treatment to 90 days.
Population: Eligible patients who began study treatment.
Measure: Number; unit: participants
Arm/Group | Treatment (Radiation Therapy, Bevacizumab, Cisplatin)
Number analyzed (Participants) | 49
participants
  Serious Adverse Events | 0
  Adverse Events | 15
Statistical Analysis 1: Comparison: Treatment (Radiation Therapy, Bevacizumab, Cisplatin); Test type: Other; Based on a report by Laciano, et al. an SAE rate of 5% and AE rate of 35% were considered tolerable and an SAE rate >=20% and AE rate >=55% excessive. If there were >=6 pts with SAES or >=22 pts with AEs then the treatment would be rejected. This study design provides alpha of 0.05 and power of 90%

2. Secondary Outcome: Number of Subjects With Treatment-related SAEs and AEs as Assessed by CTCAE v. 3.0 Criteria at Any Time.
Description: Adverse events (AEs) graded using CTCAE v3.0. Grade (Gr) refers to the severity of the AE and assigns Gr 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: 1= Mild AE, 2= Moderate AE, 3= Severe AE, 4= Life-threatening or disabling AE, 5= Death related to AE. Treatment-related SAEs defined as Gr >= 4 vaginal bleeding, Gr >=4 thrombotic event, Gr >=3 arterial event, gastrointestinal (GI) bleeding , or bowel/bladder perforation, and any Gr 5 treatment-related AE. Treatment-related AEs defined as all SAEs, Gr 3-4 nausea, vomiting, or diarrhea persisting for >2 weeks despite medical intervention, Gr 4 neutropenia or leukopenia persisting for >7 days, febrile neutropenia defined as a temperature >38.5 degree Celsius and granulocytes < 1000/mm3, Grade 3-4 hematologic toxicity with the exception of neutropenia and leukopenia, and Grade 3-4 GI, renal, cardiac, pulmonary, hepatic, or neurologic AEs.
Time Frame: From start of treatment to last follow-up, up to 6.0 years. Analysis occurred after all patients had been on study for at least 2 years.
Population: Eligible patients who started study treatment
Measure: Number; unit: participants
Arm/Group | Treatment (Radiation Therapy, Bevacizumab, Cisplatin)
Number analyzed (Participants) | 49
participants
  Serious Adverse Events | 0
  Adverse Events | 18

3. Secondary Outcome: Disease-free Survival (Three-year Rate Reported)
Description: Failure is defined as local, regional, or distant disease, or death due to any cause. Disease-free survival time is defined as time from registration to the date of failure and disease-free survival rates are estimated by the Kaplan-Meier method. Patients last known to be alive and disease-free are censored at the date of last contact.
Time Frame: From registration to 3 years
Population: Eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Radiation Therapy, Bevacizumab, Cisplatin)
Number analyzed (Participants) | 49
percentage of participants | 68.7 [53.5 to 79.8]

4. Secondary Outcome: Overall Survival (Three-year Rate Reported)
Description: Overall survival time is defined as time from registration to the date of death from any cause and is estimated by the Kaplan-Meier method. Patients last known to be alive are censored at the date of last contact.
Time Frame: From registration to 3 years
Population: Eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Radiation Therapy, Bevacizumab, Cisplatin)
Number analyzed (Participants) | 49
percentage of participants | 81.3 [67.2 to 89.8]

ADVERSE EVENTS:
Description: Per the protocol, toxicity data was collected via Common Terminology Criteria (CTC) 3.0 then mapped to CTCAE 4.0 for reporting on this website. Subjects experiencing more than one of a given AE are counted only once for that AE.
Groups:
- Treatment (Radiation Therapy, Bevacizumab, Cisplatin): Patients undergo pelvic EBRT once daily, 5 days a week, for 5 weeks for a total of 45 Gy.
  Some patients also undergo low-dose rate brachytherapy twice, 1-3 weeks apart, beginning >= 4 weeks after initiating EBRT or high-dose rate brachytherapy 5 times, >= 48 hours apart, beginning >= 2 weeks after initiating EBRT. EBRT and chemotherapy are halted on the day of high-dose rate brachytherapy. Patients receive bevacizumab IV over 30-90 minutes on days 1, 15, and 29 and cisplatin IV over 60 minutes on days 1, 8, 15, 22, 29, and 35.
  Data is reported for all patients who received study treatment, which is 59 patients.
Arm/Group | Treatment (Radiation Therapy, Bevacizumab, Cisplatin)
Serious Adverse Events (participants affected / at risk) | 13/59
Other Adverse Events (participants affected / at risk) | 59/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Radiation Therapy, Bevacizumab, Cisplatin) (N=59)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Proctitis (Gastrointestinal disorders) | 1
Rectal pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Fever (General disorders) | 1
Allergic reaction (Immune system disorders) | 1
Bladder infection (Infections and infestations) | 1
Catheter related infection (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Vascular access complication (Injury, poisoning and procedural complications) | 1
GGT increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 2
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 2
White blood cell decreased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Syncope (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Thromboembolic event (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Radiation Therapy, Bevacizumab, Cisplatin) (N=59)
Anemia (Blood and lymphatic system disorders) | 32
Hearing impaired (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 4
Blurred vision (Eye disorders) | 1
Extraocular muscle paresis (Eye disorders) | 1
Flashing lights (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 11
Anal fistula (Gastrointestinal disorders) | 1
Anal pain (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 17
Diarrhea (Gastrointestinal disorders) | 30
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 4
Dysphagia (Gastrointestinal disorders) | 2
Esophagitis (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 2
Hemorrhoids (Gastrointestinal disorders) | 3
Mucositis oral (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 32
Proctitis (Gastrointestinal disorders) | 4
Rectal hemorrhage (Gastrointestinal disorders) | 5
Rectal pain (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 15
Chills (General disorders) | 4
Edema limbs (General disorders) | 4
Fatigue (General disorders) | 34
Fever (General disorders) | 4
General disorders and administration site conditions - Other (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 4
Infections and infestations - Other (Infections and infestations) | 4
Sinusitis (Infections and infestations) | 1
Soft tissue infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 3
Vaginal infection (Infections and infestations) | 3
Dermatitis radiation (Injury, poisoning and procedural complications) | 6
Ureteric anastomotic leak (Injury, poisoning and procedural complications) | 1
Activated partial thromboplastin time prolonged (Investigations) | 2
Alanine aminotransferase increased (Investigations) | 8
Alkaline phosphatase increased (Investigations) | 5
Aspartate aminotransferase increased (Investigations) | 5
Blood bilirubin increased (Investigations) | 1
Cholesterol high (Investigations) | 1
Creatinine increased (Investigations) | 5
Investigations - Other (Investigations) | 3
Lymphocyte count decreased (Investigations) | 17
Neutrophil count decreased (Investigations) | 17
Platelet count decreased (Investigations) | 26
Weight gain (Investigations) | 3
Weight loss (Investigations) | 8
White blood cell decreased (Investigations) | 41
Acidosis (Metabolism and nutrition disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 11
Dehydration (Metabolism and nutrition disorders) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 7
Hyperglycemia (Metabolism and nutrition disorders) | 17
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypernatremia (Metabolism and nutrition disorders) | 1
Hyperuricemia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 13
Hypocalcemia (Metabolism and nutrition disorders) | 11
Hypoglycemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 17
Hypomagnesemia (Metabolism and nutrition disorders) | 23
Hyponatremia (Metabolism and nutrition disorders) | 16
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 5
Dysgeusia (Nervous system disorders) | 5
Facial nerve disorder (Nervous system disorders) | 1
Headache (Nervous system disorders) | 12
Nervous system disorders - Other (Nervous system disorders) | 3
Peripheral motor neuropathy (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 5
Agitation (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 8
Depression (Psychiatric disorders) | 8
Insomnia (Psychiatric disorders) | 8
Bladder spasm (Renal and urinary disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 1
Cystitis noninfective (Renal and urinary disorders) | 5
Hemoglobinuria (Renal and urinary disorders) | 2
Proteinuria (Renal and urinary disorders) | 1
Renal and urinary disorders - Other (Renal and urinary disorders) | 3
Urinary frequency (Renal and urinary disorders) | 8
Urinary incontinence (Renal and urinary disorders) | 3
Urinary retention (Renal and urinary disorders) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
Urinary tract pain (Renal and urinary disorders) | 4
Irregular menstruation (Reproductive system and breast disorders) | 4
Lactation disorder (Reproductive system and breast disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 11
Perineal pain (Reproductive system and breast disorders) | 3
Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 1
Uterine hemorrhage (Reproductive system and breast disorders) | 1
Uterine obstruction (Reproductive system and breast disorders) | 1
Uterine pain (Reproductive system and breast disorders) | 2
Vaginal discharge (Reproductive system and breast disorders) | 11
Vaginal dryness (Reproductive system and breast disorders) | 1
Vaginal fistula (Reproductive system and breast disorders) | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 25
Vaginal inflammation (Reproductive system and breast disorders) | 5
Vaginal obstruction (Reproductive system and breast disorders) | 6
Vaginal pain (Reproductive system and breast disorders) | 4
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 5
Alopecia (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 2
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1
Skin induration (Skin and subcutaneous tissue disorders) | 2
Skin ulceration (Skin and subcutaneous tissue disorders) | 1
Telangiectasia (Skin and subcutaneous tissue disorders) | 2
Flushing (Vascular disorders) | 1
Hot flashes (Vascular disorders) | 14
Hypertension (Vascular disorders) | 6
Hypotension (Vascular disorders) | 5
Vascular disorders - Other (Vascular disorders) | 2

LIMITATIONS AND CAVEATS:
Ineligible patients are included in the adverse event reporting on ClinicalTrials.gov, but not in endpoint results, nor in any publications, per the protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less